CLINICAL TRIAL: NCT00072098
Title: Phase I Trial Of Adenoviral Vector Delivery Of The Human Interleukin-12 cDNA By Intratumoral Injection In Patients With Metastatic Colorectal Cancer To The Liver
Brief Title: Interleukin-12 Gene in Treating Patients With Liver Metastases Secondary to Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: limited funding
Sponsor: Max Sung (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Max Sung, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 97-0564; MTS-GCO-975642; MTS-GCO-971592; CDR0000335463; NIH 9911-359
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; liver metastases; recurrent rectal cancer; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Group (Experimental): Direct intratumoral injection of metastatic hepatic tumors using an adenoviral vector expressing the human recombinant interleukin-12 gene
  Interventions: Biological: adenovirus vector; Biological: interleukin-12 gene

INTERVENTIONS:
Biological: adenovirus vector
Biological: interleukin-12 gene

SUMMARY:
RATIONALE: Inserting the interleukin-12 gene into a person's cancer cells may make the body build an immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of interleukin-12 gene when injected into the tumors of patients with liver metastases secondary to colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and maximum tolerated dose of intratumoral adenoviral vector-delivered interleukin-12 gene in patients with liver metastases secondary to colorectal cancer .
* Determine the tumor response in patients treated with this regimen.
* Determine the immune response in patients treated with this regimen.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed* colorectal adenocarcinoma metastatic to the liver

  * Solitary or multiple metastatic tumors in the liver

    * Metastatic involvement of the liver no greater than 40% of estimated liver volume NOTE: *Must be from the hepatic tumor designated for study injection
* Metastatic liver tumors must be bidimensionally measurable by CT scan or MRI
* At least 1 metastatic liver tumor measuring at least 2.0 cm must be visualized by ultrasound (US) and accessible for US-guided percutaneous injection
* Extrahepatic metastases allowed
* No prior or current ascites
* Ineligible for hepatic resection

PATIENT CHARACTERISTICS:

Age

* Adult

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 16 weeks

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Hemoglobin at least 9.0 g/dL
* Platelet count at least 100,000/mm^3

Hepatic

* No clinical evidence of other severe liver disease (e.g., portosystemic encephalopathy)
* PT no greater than 14 seconds
* Bilirubin no greater than 2.0 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 45 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception during and for at least 2 months after study participation
* HIV negative
* No active infection
* No other concurrent serious medical illness
* No other malignancy within the past 5 years except inactive nonmelanoma skin cancer, carcinoma in situ of the cervix, or grade 1 papillary bladder cancer
* Oriented and rational
* Weight at least 30 kg

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy

* At least 2 months since prior corticosteroids

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 2 months since prior systemic immunosuppressive drugs
* No concurrent immunosuppressive drugs
* No concurrent anticoagulant therapy with heparin or warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
safety measure | up to day 57
  adverse event reporting
toxicity grading | up to day 57
  toxicity will assessed from grades 0 to 4 as per common toxicity criteria

SECONDARY OUTCOMES:
tumor response compared at four weeks to baseline | baseline and four weeks
  tumor masses enumerated and measured pre-treatment and 4 weeks after treatment and changes in the tumor calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Max W. Sung, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States